CLINICAL TRIAL: NCT04944511
Title: PD-1 Antibody Improve Mixed Chimerism in Patients With Hemophagocytic Lymphohistiocytosis After Allo-HCT
Brief Title: PD-1 Antibody Improve Mixed Chimerism
Acronym: HLH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, principal investigator, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PD-1, mixed chimerism
Record Dates: First submitted 2020-12-27; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: PD-1 Antibody; Mixed Chimerism
Keywords: Chimerism; PD-1
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: one group of HLH patients with mixed chimerism (80%-95%), PD-1 antibody will be used to improve the chimerism
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD-1 antibody for mixed chimerism (Experimental): PD-1 antibody (Toripalimab Injection) used for mixed chimerism in HLH patients after allo-HCT
  Interventions: Drug: Toripalimab Injection

INTERVENTIONS:
Drug: Toripalimab Injection — Toripalimab Injection used for mixed chimerism between 80%-95% in HLH patients. Dose: 240mg toripalimab Injection, two weeks later, the same dose will be repeated if patients have some improve in the chimeric rate.

SUMMARY:
PD-1/PD-L1 pathway play an important role in Inhibiting the function of antigen-specific CD8+T cells, thus matter a lot in immune escape. We intend to use PD-1 antibody to improve the function of lymhocyte and improve the chimerism in patients after allo-HCT.

DETAILED DESCRIPTION:
Mixed chimerism is a trouble condition after allogeneic hematopoietic cell transplantation (Allo-HCT),all targeted treatment are aimed to improve the function of lymphocyte recipient. PD-1 antibody was reported to restored the function of impaired lymphocyte. Therefore, we want to use PD-1 antibody to improve the function of lymhocyte and improve the chimerism in HLH patients after allo-HCT.

ELIGIBILITY:
Inclusion Criteria:

1. EBV-HLH according to the HLH-04 diagnostic criteria.
2. After allo-HCT, have achieved engraftment and reconstitute of hematopoiesis. have achieved full donor chimerism.
3. Withdraw immunosuppressive agent, chimeric rate was 80%-95%
4. Age >18 years old, gender is not limited.
5. no graft-versus-host disease was observed.
6. No secondary graft failure (ANC <0.5*10^9/l,PLT <10*10^9/l)
7. Before the start of the study, aminopherase (ALT/AST) and total bilirubin were normal. Serum creatinine ≤ 1.5 times the upper limit of Normal (ULN); No thyroid dysfunction. The left ventricular ejection fraction (LVEF) was normal.
8. Informed consent.

Exclusion Criteria:

1. Allergic to the test drug ingredients or to a more severe allergic constitution.
2. Chimeric rate continue to decline after 2 weeks of toripalimab Injection used.
3. Serious immunoreaction: myocardial damage, hepatitis, pneumonia.
4. Central nervous system symptoms.
5. Serious mental illness.
6. Active bleeding of the internal organs
7. Uncontrollable infection；
8. Pancreatitis history. Patients unable to comply during the trial and/or follow-up phase;
9. Participate in other clinical research at the same time.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Chimeric rate | 4 weeks after toripalimab injection was used
  Chimeric rate in bone marrow or peripheral blood of HLH patients

SECONDARY OUTCOMES:
treatment-related adverse events as assessed by CTCAE v5.0； | every 2 weeks after intervention, until 8 weeks after the use of PD-1 antibody
  Adverse events including thyroid function，liver function damage, myelosuppression, infection, bleeding and so on.

OTHER OUTCOMES:
Survival | 1 year
  From enrollment until death or the end of the experiment

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No